CLINICAL TRIAL: NCT07368062
Title: Study Evaluating Dexmedetomidine in the Acute Treatment of Electrical Storm: Outpatient Follow-up of Mental Health INDices (SDATE OF MIND)
Brief Title: Mental Health After Dexmedetomidine for Electrical Storm
Status: Recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 20250008-01H
Record Dates: First submitted 2025-06-03; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-05

CONDITIONS: Mental Health
Keywords: Electrical storm; Ventricular tachycardia; Dexmedetomidine; Mental health
MeSH Terms: conditions — Psychological Well-Being; Tachycardia, Ventricular | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dexmedetomidine: Treatment with dexmedetomidine during electrical storm admission
  Interventions: Drug: Dexmedetomidine
- Placebo: Usual standard of care (not including dexmedetomidine) during electrical storm admission
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion during ICU admission for electrical storm
  Groups: Dexmedetomidine
Drug: Placebo — Placebo (standard of care, no dexmedetomidine), for treatment of electrical storm while admitted to ICU
  Groups: Placebo

SUMMARY:
The goal of the research study is to measure mental health and quality of life indices of individuals treated for electrical storm (ES). The consequences of being admitted to an intensive care unit (ICU) with electrical storm as well as the treatments patients would have received, are currently not well understood. Understanding the mental health burden of these treatments among survivors can provide insights into how to improve care.

This is a study consisting of patients who participated in the SEDATE trial (dexmedetomidine vs usual standard of care to treat ES in the ICU). Patients who consent to participate in this study will be asked to complete a set of questionnaires 3-6 months after their ICU admission. The purpose of the questionnaires is to measure indices of mental health and health-related quality of life. Each questionnaire will take about 5-15 minutes to complete.

If patients have a scheduled follow-up at the University of Ottawa Heart Institute, a member of the research team will meet with them during their clinic visit to complete the questionnaires. Otherwise, they can be completed over the telephone.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an intensive care unit with a diagnosis of electrical storm within the preceding 6 months
* Previous participants in the SEDATE trial (NCT06281977)

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously admitted at the University of Ottawa Heart Institute's Intensive Cardiac Care Unit with electrical storm and enrolled in the SEDATE trial at that time will be contacted to obtain consent for study participation
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic stress disorder symptoms | Assessed 3-6 months after hospitalization for electrical storm
  Post-traumatic stress disorder (PTSD) checklist (PCL-5) score. Respondents are asked to rate the presence and severity of various symptoms in the preceding month on 5-point Likert scale. A higher score indicates worse symptoms. A cumulative cut-off score of 31-33 is usually considered indicative of probable PTSD

SECONDARY OUTCOMES:
Anxiety symptoms | Assessed 3-6 months after hospitalization for electrical storm
  General Anxiety Disorder 7-item (GAD-7). This is a screening tool for the presence and measure of the severity of anxiety symptoms. A higher score suggests more severe symptoms
Depression symptoms | Assessed 3-6 months after hospitalization for electrical storm
  Patient Health Questionnaire-9 (PHQ-9). This is a screening tool for the presence and measure of the severity of depression symptoms. A higher score suggests more severe symptoms.
Anxiety/fear relating to implantable cardioverter-defibrillator shocks | Assessed 3-6 months after hospitalization for electrical storm
  Florida Shock Anxiety Scale (FSAS). This is a measure of patient anxiety/fear relating to implantable cardioverter-defibrillator shocks. A higher score suggests more shock-related anxiety
Quality of life measure | Assessed 3-6 months after hospitalization for electrical storm
  Quality of life measurements, as obtained through use of the 36-Item Short Form Survey Instrument (SF-36), a validated questionnaire tool to measure health-related quality of life/health status across specific domains. A higher score indicates better self-reported health

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada